CLINICAL TRIAL: NCT01419392
Title: Role of Sildenafil Citrate in Patients With Unexplained Recurrent Miscarriages: a Randomized Clinical Trial
Brief Title: Role of Sildenafil Citrate in Patients With Unexplained Recurrent Miscarriages
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer El-Refaie, Lecturer of Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahmed-2004
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent Miscarriage
Keywords: sildenafil citrate; Doppler Ultrasonography; nitric oxide; total antioxidant capacity
MeSH Terms: conditions — Abortion, Habitual | interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil citrate (Experimental)
  Interventions: Drug: Sildenafil citrate
- placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Sildenafil citrate — 25 mg orally, 4 times per day for 21 days
  Other Names: Silden 25 mg tablet, EIPICO, Inc, Cairo, Egypt
  Arms: Sildenafil citrate
Drug: matching placebo — orally, 4 times per day for 21 days
  Other Names: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether sildenafil citrate is effective in improving uterine artery blood flow and oxidative stress in patients with unexplained recurrent miscarriages

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Three or more recurrent miscarriages before the 24th week of gestation with no apparent cause for their previous losses
* Three or more months have elapsed since the last abortion
* Postmenstrual period
* No other therapy allowed during our treatment course

Exclusion Criteria:

* Concomitant use of organic nitrites, or nitrates
* Severe hepatic, renal, or cardiovascular impairment
* History of stroke or myocardial infarction
* Patients with retinitis pigmentosa.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Uterine arteries blood flow | 21 days
  Uterine arteries blood flow assessed by Doppler U/S by measuring Systolic / diastolic ratio, pulsatility index and resistance index

SECONDARY OUTCOMES:
Nitric oxide serum level as a marked of oxidative stress | 21 days
Total antioxidant capacity serum level as a marker of oxidative stress | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Obstetrics and Gynecology Department, Cairo, Cairo Governorate, Egypt